CLINICAL TRIAL: NCT03206528
Title: Clinical Evaluation of the Vital Signs Monitoring System (VSMS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: G Medical Innovations Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN-7.4.7.10.20
Record Dates: First submitted 2017-06-15; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Body Temperature; Oxygen Saturation; Respiration; ECG
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- VSMS with ear unit: application of Vital Signs Monitoring System with ear unit for 6-10 days during hospitalization (throughout their admission period)
  Interventions: Device: Vital Signs Monitoring System
- VSMS without ear unit: application of Vital Signs Monitoring System without ear unit for 6-10 days during hospitalization (throughout their admission period)
  Interventions: Device: Vital Signs Monitoring System

INTERVENTIONS:
Device: Vital Signs Monitoring System — The VSMS will be adhered to each enrolled patient for the entire hospitalization period.

SUMMARY:
This is an observational, cohort-based, single-site, prospective study conducted in accordance with ISO 14155-1:2003 and ISO 14155-1:2011. The primary objectives are to evaluate the accuracy of the device's measurements/readings in comparison to a gold standard or standard of care patient monitor.

DETAILED DESCRIPTION:
This is an observational, cohort-based, single-site, prospective clinical study enrolling up to 100 patients who are hospitalized in the internal ward. There is no control group.

The primary objectives of the study are:

1. Evaluate the body temperature measured by the ear unit and validate its accuracy.
2. Evaluate the accuracy of SPO2 signals and results by comparing the readings to a gold standard device with a finger sensor.
3. Evaluate the ECG and respiration signals recorded by the patch device by comparing them to the signals recorded by a patient monitor with standard leads.

   The secondary objectives of the study are:
4. Usability - evaluate the ease of use of the device by medical staff and patients (e.g., positioning, activation, replacement of patch, understanding processes and requirements).
5. Evaluate the signals quality and the patch adherence after 5 - 7 days on the chest.

The study will assess the safety and effectiveness of the Vital Signs Monitoring System (VSMS) for its intended use/proposed indications. Data will be collected while the VSMS is adhered to each patient for the entire hospitalization period, up to 7 days. There is no follow-up required.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age above 18 years from both genders
* American Society of Anesthesiologists (ASA) physical status classification of 1-4
* Hospitalized in internal ward

Exclusion Criteria:

* Abuse of alcohol or illicit drugs
* History of mental retardation or any mental disease
* Skin irritation / Atopic dermatitis or any other skin condition in the area of patient's upper chest that might affect his/her ability to adhere the device appropriately

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients of both genders, above 18 years of age, with ASA physical status classified as 1-4. In order to obtain the necessary results, the following shall also define the patient population:
  Temperature: 30-50% of subjects shall be febrile, i.e., having:
  * An elevated core or rectal temperature of 38.0°C or higher as measured by a clinical thermometer.
  * An elevated sublingual temperature of 37.5°C or higher as measured by a clinical thermometer.
  * An elevated Axillary temperature of 37.2°C or higher as measured by a clinical thermometer.
  SPO2: 10-20% of patients shall have a blood oxygen saturation level of 70-90%.
  ECG / Respiration: At least 20% of patients shall have some type of arrhythmia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-04-25 (Actual); Primary Completion 2017-07-31 (Estimated); Study Completion 2017-07-31 (Estimated)

PRIMARY OUTCOMES:
Skin Temperature measured in units of Celsius/Fahrenheit | 6-10 days
  Validation of measurement accuracy of skin temperature as compared to gold standard.
Oxygen Saturation measured in units of percentage peripheral saturated oxygen | 6-10 days
  Validation of measurement accuracy of peripheral oxygen saturation as compared to gold standard.
.ECG signal recording and Respiration measured in units heart beat per minute | 6-10 days
  Assess quality of device's recorded ECG and respiration signals as compared to patient monitor with standard leads

SECONDARY OUTCOMES:
Quality of recorded signal | after 5-7 days of device usage
  Evaluate the quality of recorded signals in time by comparing signal of day 1 with signal in last day of adherence of the patch

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Tishler, Professor, Principal Investigator — Assaf Harofeh Hospital/Medical Center
Locations (1):
- Internal Ward B, Aliza Begin Building, Assaf Harofe Hospital (2nd Floor), P.O. Beer Ya'akov, Zerifin, Israel

IPD SHARING:
Plan to Share IPD: No